CLINICAL TRIAL: NCT06858384
Title: From Awareness to Action: Transforming Proton Pump Inhibitor Use in Ras Al Khaimah Through Education and Intervention: the RAK -PRIDE Study
Brief Title: RAK-PRIDE: Optimizing Proton Pump Inhibitor Use Through Education and Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAK Medical and Health Sciences University (Other)
Responsible Party: Principal Investigator, Syed Arman Rabbani, Professor Syed Arman Rabbani, RAK Medical and Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RAKMHSU/RES/2024-25/001
Record Dates: First submitted 2025-02-16; First posted 2025-03-05 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Proton Pump Inhibitors; Deprescribing; Inappropriate Use
Keywords: proton pump inhibitors; peptic ulcer disease; Deprescribing; pharmacist-led educational intervention; inappropriate use; RAK - PRIDE
MeSH Terms: conditions — Peptic Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmacist-Led Educational Intervention (Experimental): Physicians and patients in this arm will receive a multi-faceted pharmacist-led educational intervention. This includes evidence-based deprescribing guidelines, brochures, videos, and decision aids to promote appropriate use of PPIs and reduce unnecessary prescriptions. The intervention is delivered in four parts: educational brochures, deprescribing algorithm, patient action plans, and video-based education sessions.
  Interventions: Other: Pharmacist-Led Educational Intervention
- Control (Other): Participants in this arm will continue with their usual care without any pharmacist-led intervention during the 6-month study period. Physicians and patients will follow the standard clinical practice for PPI prescriptions.
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Other: Control (Standard treatment) — Participants in this arm will continue with their usual care without any pharmacist-led intervention during the 6-month study period. Physicians and patients will follow the standard clinical practice for PPI prescriptions. At the end of the 6-month period, the educational materials provided to the intervention group will be offered to the control group.
  Arms: Control
Other: Pharmacist-Led Educational Intervention — Physicians and patients in this arm will receive a multi-faceted pharmacist-led educational intervention. This includes evidence-based deprescribing guidelines, brochures, videos, and decision aids to promote appropriate use of PPIs and reduce unnecessary prescriptions. The intervention is delivered in four parts: educational brochures, deprescribing algorithm, patient action plans, and video-based education sessions.
  Arms: Pharmacist-Led Educational Intervention

SUMMARY:
The goal of this study is to determine if a pharmacist-led educational intervention can reduce the inappropriate use of proton pump inhibitors (PPIs) among adult patients (≥18 years) with potentially inappropriate PPI prescriptions in Ras Al Khaimah.

The main questions it aims to answer are:

* Can a pharmacist-led education program reduce unnecessary PPI use?
* Does the intervention improve patients' quality of life and reduce healthcare costs? Researchers will compare the intervention group (receiving pharmacist-led education and materials) to the usual care group to see if the intervention reduces PPI use and improves patient outcomes.

Participants will:

* Receive educational materials from pharmacists, including a patient educational brochure, PPI patient decision aid, PPI deprescribing pamphlet, and PPI patient action plan.
* Physicians involved will also receive a pharmaceutical intervention, which includes a physician educational brochure, PPI evidence-based deprescribing guideline, PPI deprescribing algorithm, and whiteboard videos on PPI deprescribing.
* Patients will be followed up for 6 months to monitor changes in PPI use, symptoms, and quality of life.

DETAILED DESCRIPTION:
The RAK-PRIDE Study aims to evaluate the impact of a pharmacist-led educational intervention on the inappropriate use of proton pump inhibitors (PPIs) among adult patients in Ras Al Khaimah. This intervention will focus on both patient education and physician guidance, promoting evidence-based deprescribing practices for PPIs.

ELIGIBILITY:
Inclusion Criteria:

Physicians will be eligible to participate if:

* They are prescribing PPIs in outpatient department of the study sites
* They have patients with potentially inappropriate PPI prescriptions

Patients will be eligible to participate if:

* They are ≥18 years
* They are presenting to out-patient departments of the study sites
* They have prescriptions of potentially inappropriate PPIs
* Their treating physicians are included in the study

Exclusion Criteria:

Physicians will be excluded if:

• They are involved in any other prescribing trial

Patients will be excluded if:

* They are unable to give informed consent, as judged by their physicians
* They have definitive indications for PPI use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who stopped or reduced the dose of PPIs | From enrollment to the end of treatment at 6 months

SECONDARY OUTCOMES:
Change in PPI dose (cummulative) | From enrollment to the end of treatment at 6 months
GERD symptom recurrence using the Gastroesophageal Reflux Disease Impact Scale (GIS) questionnaire | From enrollment to the end of treatment at 6 months
  Score Range:
  Minimum value: 9 (if all items are rated as 1, meaning "Never") Maximum value: 36 (if all items are rated as 4, meaning "Daily")
  Interpretation:
  A higher GIS score reflects more severe GERD symptoms and a greater negative impact on the patient's daily life.
  A lower GIS score suggests fewer or less severe GERD symptoms and a better quality of life.
Number of Medications | From enrollment to the end of treatment at 6 months
Quality of life by EuroQol 5-Dimension 5-Level (EQ-5D-5L) Questionnaire | From enrollment to the end of treatment at 6 months
  The EQ-5D-5L self-report questionnaire comprised two components: the EQ-5D-5L descriptive system and the EQ Visual Analogue Scale (EQ-VAS).
  * The first part (the descriptive system) assesses health in five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Respondents select one of five levels of severity for each dimension.. Health state index scores typically range from below 0 to 1, where 0 represents a health state considered equivalent to death, and negative values indicate conditions perceived as worse than death. A score of 1 reflects full health, with higher scores signifying greater health utility. These index scores are based on national or regional health preferences, meaning they may vary across different countries or regions.
  * The second component of the questionnaire is the Visual Analogue Scale (VAS). EQ-VAS (Visual Analog Scale) Score: Ranges from 0 to 100 100 = Best imaginable health 0 = Worst imaginable health
Potential adverse effects of PPI use | From enrollment to the end of treatment at 6 months
Number of Participants with Prescription of PPIs (Restart or Dose Increase) and/or Alternative Antireflux Treatments | From enrollment to the end of treatment at 6 months
  This outcome measure tracks the number of participants who either re-started or increased their PPI dose, or used alternative anti-reflux treatments (such as H2 antagonists, antacids, or prokinetic agents) over the 6-month period. The goal is to assess how many participants needed to resume or adjust their PPI therapy or opt for alternative treatments due to symptom recurrence or insufficient symptom control.
Revised Patients' Attitudes Toward Deprescribing (rPATD) questionnaire | From enrollment to the end of treatment at 6 months
  The Revised Patients' Attitudes Toward Deprescribing (rPATD) questionnaire consists of 22 questions across four subscales: Burden (5), Appropriateness (5), Concerns about Stopping (6), and Involvement (6). Each item is rated on a 5-point Likert scale (1 = Strongly Disagree to 5 = Strongly Agree), with a total score range of 22 to 110.
  Interpretation of Scores:
  A low rPATD score (closer to 22) suggests that a patient perceives their medications as necessary, has concerns about stopping them, or prefers not to be involved in deprescribing decisions.
  A high rPATD score (closer to 110) indicates that a patient feels their medications may be burdensome, sees some as unnecessary, is less concerned about stopping them, and is more open to discussing deprescribing with their healthcare provider.
Health Care Professionals' Attitudes Towards Deprescribing (HATD) Tool | From enrollment to the end of treatment at 6 months
  The Health Care Professionals' Attitudes Towards Deprescribing (HATD) tool assesses perceptions of deprescribing in older adults with limited life expectancy. It includes five domains: concerns, medication burden, organizational support, assurance, and patient involvement. Scores range from 1 to 5.
  The total HATD score is the average of five domain scores: concerns, medication burden, organizational support, assurance, and patient involvement. Each domain score is calculated by averaging the responses within that category. The minimum possible score is 1, representing minimal agreement with deprescribing-related concerns or barriers, while the maximum score is 5, indicating strong agreement with those concerns or perceptions. Interpretation of the scores can guide interventions to address barriers and improve deprescribing practices.
Healthcare Costs (Direct Medical Costs of PPI Use) | From enrollment to the end of treatment at 6 months
  Monthly PPI medication costs per patient will be calculated before and after the intervention. Costs will be aggregated at the group level to assess total expenditure changes.
  Unit of Measure: AED per patient per month.
Quality-Adjusted Life Years (QALY) Gains | From enrollment to the end of treatment at 6 months
  Health-related quality of life will be assessed using the EuroQoL EQ-5D-5L questionnaire, administered at baseline and after 6 months. EQ-5D-5L utility scores will be used to calculate QALY gains for each group.
  Unit of Measure: QALY (Quality-Adjusted Life Years)
Cost per QALY Gained (Incremental Cost-Effectiveness Ratio, ICER) | From enrollment to the end of treatment at 6 months
  The cost per QALY gained will be calculated as the difference in total healthcare costs between the intervention and control groups, divided by the difference in QALYs gained.
  Unit of Measure: AED per QALY gained.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Arman Rabbani, Principal Investigator — RAK Medical and Health Sciences University; Mohamed El-Tanani, Principal Investigator — RAK Medical and Health Sciences University; Imran Rashid Rangraze, Principal Investigator — RAK Medical and Health Sciences University; Sathvik B Sridhar, Principal Investigator — RAK Medical and Health Sciences University; Arwa Alnahdi, Principal Investigator — Ibrahim Bin Hamad Obaidullah Hospital
Locations (1):
- Ibrahim Bin Hamad Obaidullah Hospital, Ras al-Khaimah, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilsdon TD, Hendrix I, Thynne TR, Mangoni AA. Effectiveness of Interventions to Deprescribe Inappropriate Proton Pump Inhibitors in Older Adults. Drugs Aging. 2017 Apr;34(4):265-287. doi: 10.1007/s40266-017-0442-1. PMID 28220380
- [Background] Nallapeta N, Reynolds JL, Bakhai S. Deprescribing Proton Pump Inhibitors in an Academic, Primary Care Clinic: Quality Improvement Project. J Clin Gastroenterol. 2020 Nov/Dec;54(10):864-870. doi: 10.1097/MCG.0000000000001317. PMID 32091449
- [Background] Krol N, Wensing M, Haaijer-Ruskamp F, Muris JW, Numans ME, Schattenberg G, Balen J, Grol R. Patient-directed strategy to reduce prescribing for patients with dyspepsia in general practice: a randomized trial. Aliment Pharmacol Ther. 2004 Apr 15;19(8):917-22. doi: 10.1111/j.1365-2036.2004.01928.x. PMID 15080853
- [Background] Lai A, Odom A, Roskos SE, Phillips JP. Deprescribing Inappropriate Proton Pump Inhibitors in a Family Medicine Residency Practice Office. PRiMER. 2021 Nov 2;5:43. doi: 10.22454/PRiMER.2021.290175. eCollection 2021. PMID 34841218
- [Background] Pratt NL, Kalisch Ellett LM, Sluggett JK, Gadzhanova SV, Ramsay EN, Kerr M, LeBlanc VT, Barratt JD, Roughead EE. Use of proton pump inhibitors among older Australians: national quality improvement programmes have led to sustained practice change. Int J Qual Health Care. 2017 Feb 1;29(1):75-82. doi: 10.1093/intqhc/mzw138. PMID 27920248
- [Background] Clyne B, Smith SM, Hughes CM, Boland F, Cooper JA, Fahey T; OPTI-SCRIPT study team. Sustained effectiveness of a multifaceted intervention to reduce potentially inappropriate prescribing in older patients in primary care (OPTI-SCRIPT study). Implement Sci. 2016 Jun 2;11(1):79. doi: 10.1186/s13012-016-0442-2. PMID 27255504
- [Background] Reeve E, Andrews JM, Wiese MD, Hendrix I, Roberts MS, Shakib S. Feasibility of a patient-centered deprescribing process to reduce inappropriate use of proton pump inhibitors. Ann Pharmacother. 2015 Jan;49(1):29-38. doi: 10.1177/1060028014558290. Epub 2014 Nov 10. PMID 25385826
- [Background] Farrell B, Pottie K, Thompson W, Boghossian T, Pizzola L, Rashid FJ, Rojas-Fernandez C, Walsh K, Welch V, Moayyedi P. Deprescribing proton pump inhibitors: Evidence-based clinical practice guideline. Can Fam Physician. 2017 May;63(5):354-364. PMID 28500192
- [Background] Giles G, Buchan H, Hullick C, Overs M, Duggan A. What next for the Australian Atlas of Healthcare Variation series? Focusing the system on appropriate and sustainable health care. Res Health Serv Reg. 2024 Dec 19;3(1):20. doi: 10.1007/s43999-024-00056-8. PMID 39695003
- [Background] Naunton M, Peterson GM, Deeks LS, Young H, Kosari S. We have had a gutful: The need for deprescribing proton pump inhibitors. J Clin Pharm Ther. 2018 Feb;43(1):65-72. doi: 10.1111/jcpt.12613. Epub 2017 Sep 11. PMID 28895169
- [Background] Targownik LE, Fisher DA, Saini SD. AGA Clinical Practice Update on De-Prescribing of Proton Pump Inhibitors: Expert Review. Gastroenterology. 2022 Apr;162(4):1334-1342. doi: 10.1053/j.gastro.2021.12.247. Epub 2022 Feb 17. PMID 35183361
- [Background] Shanika LGT, Reynolds A, Pattison S, Braund R. Proton pump inhibitor use: systematic review of global trends and practices. Eur J Clin Pharmacol. 2023 Sep;79(9):1159-1172. doi: 10.1007/s00228-023-03534-z. Epub 2023 Jul 7. PMID 37420019
- [Background] Kinoshita Y, Ishimura N, Ishihara S. Advantages and Disadvantages of Long-term Proton Pump Inhibitor Use. J Neurogastroenterol Motil. 2018 Apr 30;24(2):182-196. doi: 10.5056/jnm18001. PMID 29605975